CLINICAL TRIAL: NCT06550011
Title: A Phase 1/2a, Open-Label, Multiple-Cohort, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Intravitreal (IVT) Injection of ABI-110 (AAV2.N54- VEGF Trap) in Subjects With Neovascular (Wet) Age-Related Macular Degeneration (wAMD), Including Symptomatic Macular Polypoidal Choroidal Vasculopathy (PCV)
Brief Title: Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Intravitreal (IVT) Injection of ABI-110 (AAV2.N54-VEGF Trap) in Subjects With Neovascular (Wet) Age-Related Macular Degeneration (wAMD), Including Symptomatic Macular Polypoidal Choroidal Vasculopathy (PCV)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avirmax Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Avirmax ABI-110
Record Dates: First submitted 2024-07-25; First posted 2024-08-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neovascular (Wet) AMD

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Low Dose
  Interventions: Drug: ABI-110 Low Dose
- Dose level 2 (Experimental): Medium Dose
  Interventions: Drug: ABI-110 Medium Dose
- Dose level 3 (Experimental): High Dose
  Interventions: Drug: ABI-110 High Dose

INTERVENTIONS:
Drug: ABI-110 Low Dose — Low dose. lower than the safety factor of 10 as recommended by the FDA
  Arms: Dose level 1
Drug: ABI-110 Medium Dose — Medium dose
  Arms: Dose level 2
Drug: ABI-110 High Dose — High Dose
  Arms: Dose level 3

SUMMARY:
This will be a clinical study to assess initial safety and tolerability of IVT ABI-110 in patients diagnosed with wet macular degeneration (wAMD), including symptomatic macular PCV.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, multiple-cohort, dose-escalation study to evaluate the safety, tolerability, and preliminary efficacy of IVT ABI-110 (AAV2.N54-VEGF-Trap) injection in subjects with wAMD), including symptomatic macular PCV.

This trial will include a screening period, confirmation of response to EYLEA (aflibercept), single administration of ABI-110, and follow-up period of 104 weeks after IVT ABI-110 injection.

ELIGIBILITY:
Key Inclusion Criteria:

* General:

  1. Must be willing and able to provide written, signed informed consent.
  2. Age: Subjects ≥ 50 and ≤ 89 years of age at the time of signing the informed consent

     Study eye:
  3. Diagnosis of wAMD, including symptomatic macular PCV, confirmed by the Central Reading Center
  4. The macular neovascularization lesion must be confirmed as determined by the Central Reading Center based on SD-OCT imaging at screening.
  5. BCVA ≤ 20/25 and ≥ 20/250 (≤ 80L and ≥ 30L ETDRS letters)
  6. History of ≥ 2 anti-VEGF injections prior to trial entry with meaningful response to anti-VEGF and continued need for anti-VEGF treatment
  7. Response to anti-VEGF at trial entry

Key Exclusion Criteria:

* Study or Fellow Eye:

  1. Prior gene therapy, either eye
  2. Any active ocular/intraocular infection or inflammation (e.g., blepharitis, infectious conjunctivitis, keratitis, scleritis, uveitis) or history of idiopathic or autoimmune-associated uveitis, either eye
  3. History of retinal disease other than wAMD or PCV, study eye
  4. Any condition preventing visual acuity improvement (e.g., fibrosis, atrophy, or retinal epithelial tear in the center of the fovea), study eye.
  5. History of (or active) retinal detachment, study eye
  6. Uncontrolled glaucoma (defined as IOP > 25 mmHg despite treatment), study eye, or history of steroid-response ocular hypertension/glaucoma in either eye
  7. History of intravitreal therapy, (other than anti-VEGF therapy) such as intravitreal steroid injection or investigational product, in the 6 months prior to screening, study eye
  8. Any prior treatment with photodynamic therapy or laser photocoagulation, study eye
  9. History of glaucoma filtration, vitrectomy, or other procedure that could affect drug distribution or clearance, study eye.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 52 weeks
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Preliminary Efficacy | 52 weeks
  Change from baseline to Week 52 after ABI-110 treatment in BCVA as assessed by ETDRS chart at a starting distance of 4M
Pharmacokinetics and Pharmacodynamics | 52 weeks
  Changes in PK and PD by ABI-110 dose level
Immunogenicity | 52 weeks
  Changes in Anti-AAV2 antibodies (ADA) and anti-VEGF-Trap antibodies in serum
Optimal Dose | 52 weeks
  To determine the optimal dose of IVT ABI-110 injection for later phases of study

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Retina Consultants, Bakersfield, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Texas - San Antonio, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No